CLINICAL TRIAL: NCT03512483
Title: The Virtual Atrial Fibrillation Clinic: Improving Specialty Care Delivery
Brief Title: VCH -- vAFC Phase 3
Acronym: vAFC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Interior Health (Industry)
Responsible Party: Principal Investigator, Kathy Rush, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H19-03601
Record Dates: First submitted 2018-03-28; First posted 2018-04-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Cardiac; Telehealth; Older Adults
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Control group participants will be notified of their assignment and will continue their usual care with the AF clinic receiving onsite care. Participants will be contacted at 3 time points (baseline, 3 months, and 6 months)
- Virtual Atrial Fibrillation Clinic (Experimental): Participants in the intervention group can expect to receive between 1 and 4 telehealth appointments over a 6 month period, as well as being contacted by the research team at 3 time points for data collection (baseline, 3 months, and 6 months). Telehealth appointments will consist of remote interactions with clinicians. Telehealth appointments will take place in participants' homes, using their personal computer/tablet/smartphone. Participants will also receive an orientation to the website and will be encouraged to visit often and utilize the resources. To promote and encourage website interaction, emails will be sent to participants once semi-monthly for the duration of the intervention with highlights and important messages from the website.
  Interventions: Behavioral: Virtual Atrial Fibrillation Clinic

INTERVENTIONS:
Behavioral: Virtual Atrial Fibrillation Clinic — Participants in the intervention group will receive usual GP care plus the vAFC which consists of telehealth appointments with Nurse Practitioner/Cardiologist and access to an AF specific educational website. It is anticipated the vAFC, as with the onsite clinic, will include a maximum of four scheduled telehealth appointments: an initial appointment following randomization, at 4-6 weeks, 3 months, and 6 months.
  Arms: Virtual Atrial Fibrillation Clinic

SUMMARY:
The purpose of this third phase of a three-phase study is to pilot a virtual AF clinic (vAFC) compared to usual onsite care provided by a specialty AF clinic. Older adults with AF will be recruited and randomized into either the vAFC (videoconference appointments with specialists at the Vancouver AF clinic, supplemented with educational content on an AF website developed from phase one results) or the usual care group (onsite appointments with specialists at the Vancouver AF clinic). This pilot will generate evidence to determine the feasibility of scaling up the vAFC model to other sites.

DETAILED DESCRIPTION:
Background: Specialty atrial fibrillation (AF) clinics have been shown to reduce AF-related hospitalizations, emergency department readmissions, and overall healthcare costs, while at the same time improving health behaviours and quality of life for patients. An AF clinic delivered virtually may offer a viable approach to remove barriers to accessing specialty care, but currently, no virtual AF models exist. However, virtual clinics that use new and emerging digital and communications technologies have been used in managing patients with a variety of chronic diseases: inflammatory bowel disease, diabetes, kidney disease, ophthalmology problems, and for post-operative follow-up (e.g., orthopedic surgery). They have been found to facilitate rapid referral, improve communication with providers, improve clinical indicators, improve self-efficacy, and achieve knowledge comparable to usual care. Purpose: The primary purpose of phase 3 of the project is to implement and evaluate an alternative model of care, a Virtual AF Clinic (vAFC) to referred patients with AF living in communities outside the Greater Vancouver area.

Methodology:

Design: We will test two modes of AF care: 1) virtual AF care (intervention group) and 2) in person AF clinic care (control group). The intervention group will receive the vAFC. The vAFC will include up to four scheduled encounters with the NPs/cardiologist: an initial encounter following baseline work-up (e.g., Holter, echo) and at 4 to 6 weeks, 3 months, and 6 months. For the duration of the intervention, the vAFC group will also receive access to a website with specific AF educational content and resources. The control group will receive usual onsite AF care provided by the Vancouver AF clinic. Recruitment: A total of 60-80 patients with AF, 30-40 allocated to each group, will be recruited from the Vancouver AF clinic. This sample size is consistent with recommendations for pilot/feasibility studies. AF clinic staff will identify eligible patients, and will send them a "letter of initial contact" letter. Patients will contact or be contacted by the research team who will provide additional study details, answer questions, conduct screening for eligibility, and obtain consent. Data Collection: Intervention and control groups will complete the same repeated measures during the study period. Demographics will be obtained at baseline. The primary outcomes: AF

Knowledge and AF Quality of Life, and secondary outcomes:

Healthcare Utilization, and Perceived Stress, will be obtained at three time points: baseline (t1) (following consent, prior to randomization), 3 months (t2), and 6 months (t3).The secondary outcomes: Lifestyle Behaviors, Physical Activity, and Patient Satisfaction will be obtained at t1 and t3. Questionnaire data will be collected using the online survey program Qualtrics. Each participant will be assigned a unique identifier code and emailed a link to the survey and consent form once they have completed eligibility screening. Patient health history, stroke risk, bleeding risk, and medications will be extracted from the consult letter sent to the AF clinic during patient referral. Website usage will be measured for each participant using Google Analytics. Following the study, approximately eight participants from each study arm will be invited to participate in an hour-long interview. Data Analysis: The focus of the pilot will be on effect sizes, as a

guide for determining the number of cases required for a full- scale study and the feasibility for such a study. The data will be

evaluated both graphically and statistically, with an emphasis on the effect sizes of the changes across time and on the effect sizes for the group differences.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older;
* Patients with a diagnosis of atrial fibrillation confirmed through an ECG;
* first time patient at the AF Vancouver clinic;
* live outside Vancouver city;
* have no problems with memory and recall;
* will be English speaking or have a family member who can assist with reading, understanding and completing the consent and survey documents;
* able to give own consent to participate in this study;
* have access to a computer/tablet/laptop with reliable internet;
* participate voluntarily and freely.

Exclusion Criteria:

* if the participant seems like a poor candidate for virtual care based on the discretion of the AF clinic staff;
* cognitive impairment;
* uncompensated hearing impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Atrial Fibrillation Effect on Quality of Life (AFEQT) | baseline, 3 months and 6 months
  Atrial Fibrillation Effect on QualiTy-of-Life Questionnaire (AFEQT), a 20 item, 7-point scale, with four domains: Symptoms, Daily Activities, Treatment Concerns, and Satisfaction.
Change from baseline Atrial Fibrillation Knowledge | baseline, 3 months and 6 months
  Multiple choice survey with three response options, asking questions about atrial fibrillation, including questions regarding symptoms, treatment, medications, risk factors, and lifestyle.

SECONDARY OUTCOMES:
Healthcare Utilization | baseline, 3 months and 6 months
  patient documentation of all health encounters related to their atrial fibrillation, who initiated the encounter, date, and result of encounter, as well as any indirect costs.
Perceived Stress | baseline, 3 months and 6 months
  The Perceived Stress Scale (PSS-14), a 14-item, 5-point scale, will measure the degree to which situations in ones life are considered stressful, ability to control aspects of life, confidence in handling problems, or being unable to cope with demands.
Smoking behaviour | baseline and 6 months
  Two questions determining whether the participant uses tobacco products, and if yes, how often in the past month they use those tobacco products.
Alcohol consumption | baseline and 6 months
  Three questions determining whether participants drink alcohol, how often they drink alcohol, and how much alcohol they drink.
Nutrition | baseline and 6 months
  Five questions determining in a "typical week" how many days participants eat fruit and vegetables, how many servings of fruit and vegetables they eat, and what type of fat or oil is used in food preparation.
Physical Activity | baseline and 6 months
  Phone Frequency Intensity Time Type (FITT) Questionnaire - measuring often, how long, how out of breath, and what kinds of physical activity have been performed in a typical week.
Waist Circumference | baseline and 6 months
  Waist circumference in centimeters recorded at the top of the Iliac crest.
Weight | baseline and 6 months
  Weight in kilograms or pounds. Used in the calculation of Body Mass Index.
Height | baseline and 6 months
  Height in meters or feet. Used in the calculation of Body Mass Index.
Bleeding Risk | baseline and 6 months
  HAS-BLED tool to assess bleeding risk includes 7 risk factors, and a score equal to or greater than 3 indicates high risk of bleeding.
Stroke Risk | baseline and 6 months
  CHA2DS2-VASc to assess risk of stroke includes 8 parameters assigned 1-2 points for a total score of 10; scores reflect need for anticoagulation.
Website Usage | baseline to 6 months
  Using Google Analytics, participant website usage will include time spent on the website, number of visits, pages visited, page scroll depth, videos watched, content downloaded, external links clicked, as well as dates and times of website visits.
Demographics and health history | baseline
  Patient demographics and health history including Age, sex, date of AF diagnosis, treatments since diagnosis, AF type, cardiac risk factors, co-morbidities, medication profile and history.
Patient satisfaction | 6 months
  A modified version of the EUPS-AF will collect patient access to information; ease of health care, general assessment of healthcare provision, use of prescription medications, and relationship with care providers

CONTACTS AND LOCATIONS:
Overall Officials: Kathy L Rush, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada